CLINICAL TRIAL: NCT00107042
Title: Hepatitis B Vaccination in Youth at Adolescent Trial Network Sites: Effectiveness of Two Strategies and Evaluation of Tools To be Used in Future HIV Prevention Trials.
Brief Title: Effectiveness of Two Hepatitis B Vaccines in HIV-negative Youths
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ATN 025
Record Dates: First submitted 2005-04-04; First posted 2005-04-05 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2016-03

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HIV vaccine trial
MeSH Terms: conditions — Hepatitis B | interventions — Recombivax HB; twinrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants receive doses of Recombivax at weeks 0 and 24. A risk-behavior assessment is administered at week 12 and post-vaccination follow-up visits and bloodwork occur at weeks 28 and 76.
  Interventions: Biological: Recombivax
- 2 (Experimental): Participants receive doses of Twinrix at weeks 0 and 24. A risk-behavior assessment is administered at week 12 and post-vaccination follow-up visits and bloodwork occur at weeks 28 and 76.
  Interventions: Biological: Twinrix

INTERVENTIONS:
Biological: Recombivax — Participants receive doses of Recombivax at weeks 0 and 24.
  Arms: 1
Biological: Twinrix — Participants receive doses of Twinrix at weeks 0 and 24.
  Arms: 2

SUMMARY:
This study will evaluate 2 licensed vaccine products (Recombivax and Twinrix) given in a two-dose schedule to youth at risk for hepatitis B and HIV infection to evaluate immunogenicity of the products in this population, barriers to vaccine delivery, and factors which predict a diminished immune response. Since these youths are also potential candidates for future HIV vaccine trials, this study will also include preliminary assessment of youths' understanding of informed consent forms, and willingness to participate in a vaccine trial and return for multiple visits (including blood draws for immunologic assessment).

DETAILED DESCRIPTION:
Hepatitis B (HBV) prophylactic immunization has been recommended for at-risk adolescents for more than 10 years although universal coverage has not been achieved. Vaccine response in healthy adolescents has generally been reported to be excellent. But, data from the study Reaching for Excellence in Adolescent Care and Health (REACH) that studied HIV-negative adolescents who were at-risk of acquiring Hepatitis B infection through sexual or needle sharing behaviors has demonstrated a much lower than expected vaccine response rate in this population using standard vaccine dosing. Some data suggest that factors such as gender or body mass index might be responsible for the differences in response to the vaccine observed in individuals. The reason for the diminished vaccine response in this population is unclear. If in fact, Hepatitis B vaccine response is diminished in this population, then efforts to determine correlates of response and to improve the response are warranted. The proposed trial will evaluate 2 licensed vaccine products given in a two-dose schedule in youth at risk for hepatitis B and HIV infection to evaluate immunogenicity of the products in this population, barriers to vaccine delivery, and factors which predict a diminished immune response.

Since these youths are also potential candidates for future HIV vaccine trials, participation in such trials will require ability to understand and willingness to volunteer for such trials, ability to return for multiple vaccinations and blood draws to assess vaccine response, and willingness to participate in HIV prevention education. A hepatitis B vaccine trial will provide a licensed vaccine to youth in whom the vaccine is indicated and will allow preliminary assessment of youth's willingness to participate in a vaccine trial that involves blood draws for immunologic assessment.

Tools that will be necessary for HIV vaccine trials in youth include a youth-friendly simplified vaccine trial education component with a required written test for the participant, a standardized risk reduction education program, and a computer-assisted assessment of youth behaviors. These tools can be finalized and field tested in youth participating in the hepatitis B vaccine trial without promoting a false sense of protection from HIV. Secondary objectives of this trial will include assessment of a number of ancillary tools crucial for future HIV vaccine trials. This Hepatitis B vaccine trial will also serve as a HIV vaccine preparedness trial for youth at risk for both Hepatitis B and HIV.

Design: This is a phase II, randomized, single-blinded trial of two hepatitis B immunization regimens in 150 HIV-negative, hepatitis B core antibody, hepatitis B surface antigen and surface antibody negative youth. Vaccinations will be given in a two-dose regimen at 0 and six months (75 subjects in each arm) and the primary outcome will be seroresponsiveness one month after the 6-month dose. Safety and tolerability will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative youth age 12-17 years (No serologic evidence of HIV infection).
* Negative hepatitis B serology. (No serologic evidence of hepatitis B surface antigen (HBSAg), hepatitis B surface antibody (HBsAb or anti-HBs) and hepatitis B core antibody (HBcAb or anti-HBc)).
* Either no prior hepatitis B immunizations or unknown or incomplete hepatitis B immunization status.
* Willing to participate in HIV risk-reduction counseling and computer assisted measurement of behaviors.
* Parent or legal guardian willing to provide written permission
* Females of childbearing potential must have a negative pregnancy test at screening and should agree to avoid pregnancy through the end of the vaccine phase of the study. Females who are engaging in sexual intercourse must be willing to practice a reliable method of birth control through the end of the vaccine-phase of the study (approximately 6 months). The decision of what is "reliable" is at the discretion of the site investigator.

Exclusion Criteria:

* Presence of any serious illness requiring treatment with systemic medications, excluding treatment for asthma.
* Previous allergic reaction to any vaccines or to constituents of these vaccines (yeast, thimerosal or aluminum)
* Pregnancy
* Current immunomodulator therapy
* Receipt of immunosuppressor therapy (more than 10 mg/day of prednisone or equivalent for >1 week) in the 6 months preceding entry or anticipated long-term corticosteroid therapy in the above dose and duration. Short term (< 7 days) steroid use for the treatment of asthma is not an exclusion.
* Receipt of any vaccine within 2 weeks preceding study entry.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2004-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleen K. Cunningham, MD, Study Chair — Duke University
Locations (11):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital National Medical Center, Washington D.C., District of Columbia
  - University of Southern Florida College of Medicine, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Montefiore Medical Center, The Bronx, New York
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- Unversity of Peurto Rico School of Medicine, San Juan, Puerto Rico

REFERENCES:
- [Derived] Cunningham CK, Rudy BJ, Xu J, Bethel J, Kapogiannis BG, Ahmad S, Wilson CM, Flynn PM; Adolescent Medicine Trials Network for HIV/AIDS Interventions. Randomized trial to determine safety and immunogenicity of two strategies for hepatitis B vaccination in healthy urban adolescents in the United States. Pediatr Infect Dis J. 2010 Jun;29(6):530-4. doi: 10.1097/INF.0b013e3181d285c7. PMID 20173677
- See also: Adolescent Trials Network for HIV/AIDS Intervention — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was started in February 2004 and was completed in July 2008. A total of 11 sites, all in the United States and Puerto Rico, participated in the study.
Groups:
- Recombivax: Active Comparator: 1st dose at Week 0, 2nd dose at Week 24
- Twinrix: Experimental: 1st dose at Week 0, 2nd dose at Week 24
Period: Overall Study
Arm/Group | Recombivax | Twinrix
Started | 60 | 63
Completed | 38 | 47
Not Completed | 22 | 16
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Moved out of area | 5 | 3
Not completed — Pregnancy | 1 | 1
Not completed — Inadvertent enrollment | 0 | 1
Not completed — vaccinated outside window | 1 | 1
Not completed — Disallowed medications | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombivax | Twinrix | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.02 (1.43) | 15.22 (1.71) | 15.12 (1.58)
Age, Customized [Number; unit: participants]
  12 - 14 years | 18 | 23 | 41
  15 - 17 years | 42 | 40 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 41 | 36 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 3 | 6 | 9
  More than one race | 37 | 43 | 80
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Seroresponsiveness to Hepatitis B Surface Antigen
Description: Seroresponsiveness to Hepatitis B Surface Antigen is defined as follows:
  Responder: serum antibody level is greater than or equal to 10 mIU/mL. Non-responder: serum antibody level is less than 10 mIU/mL.
Time Frame: Week (Wk) 28 (One month after the second immunization)
Population: Participants were included if they were vaccinated at least once (Intent-to-Treat)
Measure: Number; unit: Participants
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 47 | 55
Participants
  Responder | 41 | 52
  Non-responder | 6 | 3
Statistical Analysis 1: Comparison: Recombivax vs Twinrix; The study wasn't powered to compare the 2 arms but to detect a large difference. A quantitative antibody (a'body) response was measured, but for sample size and power considerations, the outcome was considered to be binary. The primary analysis involved straightforward computation of point estimates and exact confidence intervals of immunogenicity in each arm. The data for primary analysis used the Intent-to-Treat for subjects who were vaccinated at least once. Missing titers were not imputed; Test type: Superiority or Other; p = 0.2954, Fisher Exact
Statistical Analysis 2: Comparison: Recombivax; Two-sided confidence intervals (CI) were calculated for both the "Recombivax" and "Twinrix" arms. The CI for the "Recombivax" arm is presented here; Test type: Superiority or Other; 95% confidence interval; Response Rate = 87.23, 95% CI 2-sided [74.26 to 95.17]
Statistical Analysis 3: Comparison: Twinrix; Two-sided confidence intervals (CI) were calculated for both the "Recombivax" and "Twinrix" arms. The CI for the "'Twinrix" arm is presented here; Test type: Superiority or Other; 95% confidence interval; Response Rate = 94.55, 95% CI 2-sided [84.88 to 98.86]

2. Secondary Outcome: Quantitative Vaccine Response
Description: The Log10 titer was used as the quantitative vaccine response.
Time Frame: Week 28
Population: Subjects who had a wk 28 Hep B a'body titer and was no more than 8 wks after the 2nd vaccination were included. 1 subject was missing wk 28 titer. The a'body at week 48 was positive, so subject was treated as a responder for the binary measure. For the continuous a'body titer, the exact number could not be assumed; subject was treated as missing.
Measure: Mean (Standard Deviation); unit: Log10 titer (mIU/ml)
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 47 | 54
Log10 titer (mIU/ml) | 2.29 (0.82) | 2.58 (0.65)
Statistical Analysis 1: Comparison: Recombivax vs Twinrix; Analysis included an assessment of quantitative titer values in each of the two arms using confidence intervals and examining the frequency distributions of the titers in each arm. Transformations were considered (log10) for the titers based on the distributional properties observed in the sample, with the goal of attaining approximate normality of the transformed data; Test type: Superiority or Other; p = 0.0608, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Recombivax; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; 95% confidence interval; Mean response = 2.29, 95% CI 2-sided [2.05 to 2.53]
Statistical Analysis 3: Comparison: Twinrix; Two-sided confidence intervals (CI) were calculated for both the "Recombivax" and "Twinrix" arms. The CI for the "Twinrix" arm is presented here; Test type: Superiority or Other; 95% confidence interval; Response rate = 2.58, 95% CI 2-sided [2.40 to 2.76]

3. Primary Outcome: Safety and Tolerability of Vaccine Regimens of Recombivax and Twinrix (Number of Participants With >=1 Adverse Event (AE))
Description: Frequency Distribution of AEs by Study Arm and Preferred Term. The safety and tolerability of each vaccine was assessed by measuring reactogenicity. The reactions were coded as "Any" vs. "None". In summarizing the distribution of AEs, the number of subjects with at least one event by preferred term and study arm were reported.
Time Frame: Week 12, Week 24, Week 28, Week 76
Population: The safety and tolerability of each vaccine was assessed and reported among all enrolled participants (per-protocol) after baseline at each visit visit. The data presented are cumulative for events identified at each time point.
Measure: Number; unit: participants
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 60 | 63
participants | 6 | 4

4. Primary Outcome: Safety and Tolerability of Vaccine Regimens of Recombivax and Twinrix: Serious Adverse Events (SAE)(Number of Subjects With >= 1 SAE)
Description: Frequency Distribution of SAE by Study Arm and Preferred Term. The safety and tolerability of each vaccine was assessed by measuring reactogenicity. The reactions were coded as "Any" vs. "None". The number of participants with at least one SAE is reported.
Time Frame: Week 12, Week 24, Week 28, Week 76
Population: The safety and tolerability of each vaccine was assessed and reported among all enrolled participants (per-protocol) after baseline. The data presented are cumulative for events identified at each time point.
Measure: Number; unit: participants
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 60 | 63
participants
  Asthenia | 1 | 0
  Forearm fracture | 1 | 0
  Road traffic accident | 0 | 1
  Anxiety | 0 | 1

5. Secondary Outcome: Unadjusted Relationship of Hepatitis B Vaccine Response (Log10 Titer) and Potential Impact Factors Among Subjects Whose Week 28 Antibody Results Are Within Week 28 Visit Window.
Description: The Log10 titer at Week 28 was used as the quantitative continuous vaccine response.
Time Frame: Week 28
Population: The data for this analysis included those who had a week 28 hepatitis B antibody titer and the week 28 visit window was no more than 8 weeks after the second vaccination (as treated population).
Measure: Number; unit: Participant
Groups:
- All Participants: All participants who had a week 28 hepatitis B antibody titer and the week 28 visit window was no more than 8 weeks after the second vaccination (per protocol). Participants were vaccinated at Week 0 and Week 24 with either Recombivax or Twinrix.
Arm/Group | All Participants
Number analyzed (Participants) | 75
Participant
  Study Arm: Recombivax | 34
  Study Arm: Twinrix | 41
  Site Effect: Other Site | 43
  Site Effect: Baltimore | 32
  Age: 15 - 17 years | 51
  Age: 12 - 14 years | 24
  Gender: Female | 29
  Gender: Male | 46
  Hispanic Ethnicity: No | 23
  Hispanic Ethnicity: Yes | 52
  Racial Background: White | 6
  Racial Background: Other/Mixed Race | 47
  Racial Background: Black/African American | 22
  Tanner Stage for Females: Stage 5 | 17
  Tanner Stage for Females: Stages 1 - 4 | 12
  Tanner Stage for Males: Stage 5 | 15
  Tanner Stage for Males: Stages 1 - 4 | 31
  BMI at Baseline: Normal and Underweight (<25.0) | 49
  BMI at Baseline: Overweight and Obese (>=25.0) | 26
  Ever Smoked Cigarettes: No | 59
  Ever Smoked Cigarettes: Yes | 16
  Sexual Identity: Straight (Heterosexual) | 67
  Sexual Identity: Gay, Bi, Not Sure or Undecided | 8
  Age First Sex Not Forced: Never | 44
  Age First Sex Not Forced: <=14 Years | 8
  Age First Sex Not Forced: 15-17 Years | 17
  Total Lifetime Sex Partners: 0 Partners | 44
  Total Lifetime Sex Partners: 1-5 Partners | 19
  Total Lifetime Sex Partners: >= 6 Partners | 10
  Total Lifetime Male Sex Partners: 0 Partners | 58
  Total Lifetime Male Sex Partners: 1-5 Partners | 10
  Total Lifetime Male Sex Partners: >= 6 Partners | 5
  Total Lifetime Female Sex Partners: 0 Partners | 57
  Total Lifetime Female Sex Partners: 1-5 Partners | 11
  Total Lifetime Female Sex Partners: >= 6 Partners | 5
  Ever Drank Alcohol: No | 45
  Ever Drank Alcohol: Yes | 30
  Ever Smoked Marijuana: No | 58
  Ever Smoked Marijuana: Yes | 17
  Ever Used Drugs not Prescribed: No | 71
  Ever Used Drugs not Prescribed: Yes | 4
Statistical Analysis 1: Comparison: All Participants; This is a regression analysis for testing the effect of treatment arm (Recombivax vs. Twinrix) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.1667, Regression, Linear; Regression coefficient = 0.2455, Standard Error of Mean 0.1757
Statistical Analysis 2: Comparison: All Participants; This is a regression analysis for testing the effect of site effect(Other sites vs. Baltimore) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.9890, Regression, Linear; Regression coefficent = -0.0025, Standard Error of Mean 0.1792
Statistical Analysis 3: Comparison: All Participants; This is a regression analysis for testing the effect of age(15 - 17 year old particpants vs. 12 - 14 year old participants) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.2796, Regression, Linear; Regression coeffcient = 0.2053, Standard Error of Mean 0.1885
Statistical Analysis 4: Comparison: All Participants; This is a regression analysis for testing the effect of gender(Females vs. Males) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.0080, Regression, Linear; Regresssion coeffcient = -0.4726, Standard Error of Mean 0.1734
Statistical Analysis 5: Comparison: All Participants; This is a regression analysis for testing the effect of Hispanic ethnicity (Not Hispanic vs. Hispanic) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.2543, Regression, Linear; Regression coefficient = 0.2189, Standard Error of Mean 0.1905
Statistical Analysis 6: Comparison: All Participants; This is a regression analysis for testing the effect of racial background(White vs. Other/Mixed vs. Black/African American) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between White vs. Other/Mixed Race is presented; Test type: Superiority or Other; p = 0.3661, Regression, Linear; Regression coefficient = 0.2994, Standard Error of Mean 0.3292
Statistical Analysis 7: Comparison: All Participants; This is a regression analysis for testing the effect of racial background(White vs. Other/Mixed vs. Black/African American) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between White vs. Black/African American is presented; Test type: Superiority or Other; p = 0.9812, Regression, Linear; Regression coefficient = 0.0083, Standard Error of Mean 0.3497
Statistical Analysis 8: Comparison: All Participants; This is a regression analysis for testing the effect of Tanner Stage for Females(Stage 5 vs. Stages 1 - 4) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.7766, Regression, Linear; Regression coefficient = -0.0663, Standard Error of Mean 0.2314
Statistical Analysis 9: Comparison: All Participants; This is a regression analysis for testing the effect of Tanner Stage for Males(Stage 5 vs. Stages 1 - 4) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.2492, Regression, Linear; Regression coefficient = -0.2929, Standard Error of Mean 0.2508
Statistical Analysis 10: Comparison: All Participants; This is a regression analysis for testing the effect of BMI at Baseline(Normal and Underweight (<25.0) vs. Overweight and Obsese (>= 25.0)) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.0877, Regression, Linear; Regression coeffcient = -0.3160, Standard Error of Mean 0.1826
Statistical Analysis 11: Comparison: All Participants; This is a regression analysis for testing the effect of BMI at Baseline(continuous variable) on vaccine response as measured in log10 titers; Test type: Superiority or Other; p = 0.0117, Regression, Linear; Regression coefficient = -0.0292, Standard Error of Mean 0.0113
Statistical Analysis 12: Comparison: All Participants; This is a regression analysis for testing the effect of smokng cigarettes(Never Smoked vs. Has Smoked) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.7899, Regression, Linear; Regression coefficient = -0.0578, Standard Error of Mean 0.2163
Statistical Analysis 13: Comparison: All Participants; This is a regression analysis for testing the effect of sexual identity(Straight (heterosexual) vs. Gay (homosexual), Bi (bisexual), and Not Sure or Undecided) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.0607, Regression, Linear; Regression coefficient = -0.5339, Standard Error of Mean 0.2803
Statistical Analysis 14: Comparison: All Participants; This is a regression analysis for testing the effect of age at which the subject first had unforced sex (Never vs. <= 14 year olds vs. 15-17 year olds) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between "never" vs. "<= 14 year olds" is presented; Test type: Superiority or Other; p = 0.1670, Regression, Linear; Regression coefficient = -0.3883, Standard Error of Mean 0.2779
Statistical Analysis 15: Comparison: All Participants; This is a regression analysis for testing the effect of age at which subject had first unforced sex (Never vs. <= 14 year olds vs. 15 - 17 year olds) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between "never" vs. "15-17 year olds" is presented; Test type: Superiority or Other; p = 0.8682, Regression, Linear; Regression coefficient = 0.0344, Standard Error of Mean 0.2065
Statistical Analysis 16: Comparison: All Participants; This is a regression analysis for testing the effect of total number of lifetime sex partners (0 partners vs. 1-5 partners vs. >= 6 partners) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between 0 partners vs. 1-5 partners is presented; Test type: Superiority or Other; p = 0.4219, Regression, Linear; Regression coefficient = 0.1532, Standard Error of Mean 0.1896
Statistical Analysis 17: Comparison: All Participants; This is a regression analysis for testing the effect of Total Number of Lifetime Sex Partners(0 partners vs. 1-5 partners vs. >= 6 partners) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between 0 partners vs. >= 6 partners is presented; Test type: Superiority or Other; p = 0.0020, Regression, Linear; Regression coefficient = -0.7752, Standard Error of Mean 0.2420
Statistical Analysis 18: Comparison: All Participants; This is a regression analysis for testing the effect of Total Number of Male Lifetime Sex Partners(0 partners vs. 1-5 partners vs. >= 6 partners) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between 0 partners vs. 1-5 partners is presented; Test type: Superiority or Other; p = 0.1659, Regression, Linear; Regression coefficient = 0.2921, Standard Error of Mean 0.2086
Statistical Analysis 19: Comparison: All Participants; This is a regression analysis for testing the effect of Total Number of Male Lifetime Sex Partners(0 partners vs. 1-5 partners vs. >= 6 partners) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between 0 partners vs. >= 6 partners is presented; Test type: Superiority or Other; p = 0.0000, Regression, Linear; Regression coefficient = -1.6163, Standard Error of Mean 0.2839
Statistical Analysis 20: Comparison: All Participants; This is a regression analysis for testing the effect of Total Number of Female Lifetime Sex Partners(0 partners vs. 1-5 partners vs. >= 6 partners) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between 0 partners vs. 1-5 partners is presented; Test type: Superiority or Other; p = 0.4701, Regression, Linear; Regression coefficient = -0.1788, Standard Error of Mean 0.2463
Statistical Analysis 21: Comparison: All Participants; This is a regression analysis for testing the effect of Total Number of Female Lifetime Sex Partners(0 partners vs. 1-5 partners vs. >= 6 partners) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups. In this statistical analysis, information for the comparison between 0 partners vs. >= 6 partners is presented; Test type: Superiority or Other; p = 0.7572, Regression, Linear; Regression coefficient = 0.1083, Standard Error of Mean 0.3488
Statistical Analysis 22: Comparison: All Participants; This is a regression analysis for testing the effect of whether a subject ever drank alcohol (No vs. Yes) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.8657, Regression, Linear; Regression coefficient = -0.0307, Standard Error of Mean 0.1809
Statistical Analysis 23: Comparison: All Participants; This is a regression analysis for testing the effect of whether a subject ever smoked marijuana(No vs. Yes) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.0917, Regression, Linear; Regression coefficient = -0.3548, Standard Error of Mean 0.2076
Statistical Analysis 24: Comparison: All Participants; This is a regression analysis for testing the effect of whether a subject ever used drugs not prescribed(No vs. Yes) on vaccine response as measured in log10 titers. The null hypothesis is no difference between groups; Test type: Superiority or Other; p = 0.3788, Regression, Linear; Regression coefficient = -0.3474, Standard Error of Mean 0.3924

6. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen (Binary); Predictor: STUDY ARM.
Description: Qualitative Vaccine Response to Hepatitis B Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Study arm was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: Participants who had a Wk 28 Hep B a'body titer were included. One subject had no results at Wk 28 but had results at entry and end of study (EOS). Since the EOS titer was > 10, this subject was included as a responder in qualitative analyses, but not in quantitative analyses, since the EOS titer is not sufficiently predictive of the Wk 28 titer.
Measure: Number; unit: Participants
Groups:
- Recombivax: Active Comparator: 1st dose at Week 0, 2nd dose at Wk 24
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 47 | 55
Participants
  Responder | 41 | 52
  Non-Responder | 6 | 3
Statistical Analysis 1: Comparison: Recombivax vs Twinrix; Test type: Superiority or Other; p = 0.2068, Univariate regression, logistic; Odds Ratio (OR) = 2.54, 95% CI 2-sided [0.60 to 10.76] — The reference group is the 'Recombivax' group

7. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: SITE EFFECT
Description: Qualitative Vaccine Response to Hepatitis B Surface Antigen is defined as a "Responder" if serum antibody level is >= 10 mIU/mL and a "Non- Responder" if a serum a'body level is < 10 mIU/mL. Site effect was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Other Sites: All other clinical sites (besides the Baltimore site) where subjects were enrolled.
- Baltimore: Clinical site where subjects were enrolled.
Arm/Group | Other Sites | Baltimore
Number analyzed (Participants) | 47 | 55
Participants
  Responder | 42 | 51
  Non-Responder | 5 | 4
Statistical Analysis 1: Comparison: Other Sites vs Baltimore; Test type: Superiority or Other; p = 0.5524, Univariate regression, logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.38 to 6.01] — The reference group is the 'Other Sites' group

8. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: AGE
Description: Qualitative Vaccine Response to Hepatitis B (Hep B)Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Age was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- 15-17 Years of Age: Subjects between the ages of 15 and 17 years, inclusive
- 12-14 Years of Age: Subjects between the ages of 12 and 14 years, inclusive
Arm/Group | 15-17 Years of Age | 12-14 Years of Age
Number analyzed (Participants) | 68 | 34
Participants
  Responder | 61 | 32
  Non-Responder | 7 | 2
Statistical Analysis 1: Comparison: 15-17 Years of Age vs 12-14 Years of Age; Test type: Superiority or Other; p = 0.4646, Univariate regression, logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.36 to 9.36] — The reference group is the '15-17 year' age group

9. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: GENDER
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum a'body level is < 10 mIU/mL. Gender was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Female: Female Subjects
- Male: Male Subjects
Arm/Group | Female | Male
Number analyzed (Participants) | 38 | 64
Participants
  Responder | 36 | 57
  Non-Responder | 2 | 7
Statistical Analysis 1: Comparison: Female vs Male; Test type: Superiority or Other; p = 0.3390, Univariate regression, logistic; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.09 to 2.30] — The reference group is the 'Female' group

10. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: HISPANIC ETHNICITY
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Hispanic ethnicity was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Not Hispanic: Subjects who reported they were not of Hispanic ethnicity.
- Hispanic: Subjects who reported they were of Hispanic ethnicity.
Arm/Group | Not Hispanic | Hispanic
Number analyzed (Participants) | 27 | 75
Participants
  Responder | 21 | 72
  Non-Responder | 6 | 3
Statistical Analysis 1: Comparison: Not Hispanic vs Hispanic; Test type: Superiority or Other; p = 0.0102, Univariate regression, logistic; Odds Ratio (OR) = 6.86, 95% CI 2-sided [1.58 to 29.78] — The reference group is the 'Hispanic: NO' group
Statistical Analysis 2: Comparison: Not Hispanic vs Hispanic; Test type: Superiority or Other; p = 0.0118, Multivariate regression, logistic — Since Hispanic (no, yes) was a factor with a p-value of < 0.15 in the unadjusted univariate regression analysis, it was entered into the initial full multivariate model; Odds Ratio (OR) = 7.38, 95% CI 2-sided [1.56 to 34.95] — The reference group is the "Hispanic: NO" group

11. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: RACE
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Race was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- White: Subjects who reported their race to be white.
- Other/Mixed Race: Subjects who reported their race to be other than white, black, or of mixed race.
- Black/African American: Subjects who reported their race to be black or African American
Arm/Group | White | Other/Mixed Race | Black/African American
Number analyzed (Participants) | 9 | 68 | 25
Participants
  Responder | 8 | 66 | 19
  Non-Responder | 1 | 2 | 6
Statistical Analysis 1: Comparison: White vs Black/African American; Test type: Superiority or Other; p = 0.4241, Univariate regression, logistic; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.04 to 3.84] — The reference group is the 'White' group
Statistical Analysis 2: Comparison: White vs Other/Mixed Race; Test type: Superiority or Other; p = 0.2685, Univariate regression, logistic; Odds Ratio (OR) = 4.12, 95% CI 2-sided [0.34 to 50.76] — The reference group is the 'White' group

12. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: TANNER STAGE FOR FEMALES
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Tanner stage by gender was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: Females who had a Wk 28 Hep B a'body titer were included. One subject had no results at Wk 28 but had results at entry and end of study (EOS). Since the EOS titer was > 10, this subject was included as a responder in qualitative analyses, but not in quantitative analyses, since the EOS titer isn't sufficiently predictive of the Wk 28 titer.
Measure: Number; unit: Participants
Groups:
- Tanner Stage 5 (Females): Females who were self-assessed and categorized to Tanner Stage 5.
- Tanner Stages 1-4 (Females): Females who were self-assessed and categorized to Tanner Stages 1, 2, 3, or 4.
Arm/Group | Tanner Stage 5 (Females) | Tanner Stages 1-4 (Females)
Number analyzed (Participants) | 20 | 18
Participants
  Responder | 19 | 17
  Non-responder | 1 | 1
Statistical Analysis 1: Comparison: Tanner Stage 5 (Females) vs Tanner Stages 1-4 (Females); Test type: Superiority or Other; p = 0.9390, Univariate regression, logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.05 to 15.44] — The reference group is the 'Stage 5' group

13. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: TANNER STAGE FOR MALES
Description: as for outcome 12
Time Frame: Week 28
Population: Male participants who had a Wk 28 Hep B a'body titer were included. One subject had no results at Wk 28 but had results at entry and end of study (EOS). Since the EOS titer was > 10, this subject was included as a responder in qualitative analyses, but not in quantitative analyses, since the EOS titer isn't sufficiently predictive of Wk 28 titer.
Measure: Number; unit: Participants
Groups:
- Tanner Stage 5 (Males): Males who were self-assessed and categorized to Tanner Stage 5.
- Tanner Stages 1-4 (Males): Males who were self-assessed and categorized to Tanner Stages 1, 2, 3, or 4.
Arm/Group | Tanner Stage 5 (Males) | Tanner Stages 1-4 (Males)
Number analyzed (Participants) | 22 | 42
Participants
  Responder | 19 | 38
  Non-responder | 3 | 4
Statistical Analysis 1: Comparison: Tanner Stage 5 (Males) vs Tanner Stages 1-4 (Males); Test type: Superiority or Other; p = 0.6181, Univariate regression, logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.30 to 7.39] — The reference group is the "Stage 5" group

14. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: BMI at Baseline
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. BMI at baseline was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Normal and Underweight (< 25.0): Subjects whose BMIs were normal to < 25.0
- Overweight and Obese (>=25.0): Subjects whose BMIs were >= 25.0
Arm/Group | Normal and Underweight (< 25.0) | Overweight and Obese (>=25.0)
Number analyzed (Participants) | 66 | 36
Participants
  Responder | 62 | 31
  Non-responder | 4 | 5
Statistical Analysis 1: Comparison: Normal and Underweight (< 25.0) vs Overweight and Obese (>=25.0); Test type: Superiority or Other; p = 0.1943, Univariate regression, logistic; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.10 to 1.60] — The reference group is the "Normal and Underweight (<25.0)" group

15. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: EVER SMOKED CIGARETTES
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Whether participants ever smoked cigarettes was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Ever Smoked Cigarettes: NO: Subjects who have never smoked cigarettes
- Ever Smoked Cigarettes: YES: Subjects who have smoked cigarettes
Arm/Group | Ever Smoked Cigarettes: NO | Ever Smoked Cigarettes: YES
Number analyzed (Participants) | 82 | 19
Participants
  Responder | 76 | 16
  Non-responder | 6 | 3
Statistical Analysis 1: Comparison: Ever Smoked Cigarettes: NO vs Ever Smoked Cigarettes: YES; Test type: Superiority or Other; p = 0.2542, Univariate regression, logistic; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.10 to 1.86] — The reference group is the "Ever smoked cigarettes: NO" group

16. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: SEXUAL IDENTITY
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Sexual identity was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Straight (Heterosexual): Subjects who were straight (heterosexual)
- Gay (Homosexual), Bi (Bisexual), Not Sure or Undecided: Subjects who were either gay (homosexual), bisexual, not sure or undecided.
Arm/Group | Straight (Heterosexual) | Gay (Homosexual), Bi (Bisexual), Not Sure or Undecided
Number analyzed (Participants) | 93 | 9
Participants
  Responder | 87 | 6
  Non-responder | 6 | 3
Statistical Analysis 1: Comparison: Straight (Heterosexual) vs Gay (Homosexual), Bi (Bisexual), Not Sure or Undecided; Test type: Superiority or Other; p = 0.0161, Univariate regression, logistic; Odds Ratio (OR) = 0.14, 95% CI 2-sided [0.03 to 0.69] — The reference group is the "Straight (heterosexual)" group
Statistical Analysis 2: Comparison: Straight (Heterosexual) vs Gay (Homosexual), Bi (Bisexual), Not Sure or Undecided; Test type: Superiority or Other; p = 0.0222, Multivariate regression, logistic — Since sexual identity was a factor with a p-value of < 0.15 in the unadjusted univariate regression analysis, it was entered into the initial full multivariate model; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.02 to 0.74] — The reference group is the "Straight (heterosexual)" group

17. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: AGE AT WHICH SUBJECT FIRST HAD SEX (NOT FORCED)
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Age of participants' first unforced sexual encounter was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Never: Subjects who reported they never had anal or vaginal sex because they wanted to.
- 12-14 Years of Age: Subjects who reported they first had anal or vaginal sex because they wanted to between the ages of 12 and 14, inclusive
- 15-17 Years of Age: Subjects who reported they first had anal or vaginal sex because they wanted to between the ages of 15 and 17, inclusive
Arm/Group | Never | 12-14 Years of Age | 15-17 Years of Age
Number analyzed (Participants) | 62 | 10 | 24
Participants
  Responder | 59 | 7 | 23
  Non-responder | 3 | 3 | 1
Statistical Analysis 1: Comparison: Never vs 15-17 Years of Age; Test type: Superiority or Other; p = 0.8945, Univariate regression, logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.12 to 11.83] — The reference group is the "Never" (had sex)group
Statistical Analysis 2: Comparison: Never vs 12-14 Years of Age; Test type: Superiority or Other; p = 0.0190, Univariate regression, logistic; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.02 to 0.70] — The reference group is the "Never" (had sex) group

18. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: TOTAL LIFETIME SEX PARTNERS
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Total number of lifetime sex partners was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- 0 Sex Partners: Subjects who have never had a sex partner
- 1 - 5 Sex Partners: Subjects who have had 1 - 5 lifetime sex partners
- >= 6 Sex Partners: Subjects who have had 6 or more lifetime sex partners
Arm/Group | 0 Sex Partners | 1 - 5 Sex Partners | >= 6 Sex Partners
Number analyzed (Participants) | 62 | 26 | 12
Participants
  Responder | 59 | 26 | 7
  Non-responder | 3 | 0 | 5
Statistical Analysis 1: Comparison: 0 Sex Partners vs >= 6 Sex Partners; Test type: Superiority or Other; p = 0.0042, Univariate regression, logistic; Odds Ratio (OR) = 0.08, 95% CI 2-sided [0.01 to 0.48] — The reference group is the "0 partners" group
Statistical Analysis 2: Comparison: 0 Sex Partners vs 1 - 5 Sex Partners; Test type: Superiority or Other; p = 0.6893, Univariate regression, Logistic; Odds Ratio (OR) = 1.65 — The reference group is the "0 partners" group. Two sided 95% confidence interval: Lower Limit = 0.17; upper limit = infinity

19. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: TOTAL LIFETIME MALE SEX PARTNERS
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Total number of lifetime male sex partners was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- 0 Male Sex Partners: Male and female subjects who have never had a male sex partner
- 1-5 Male Sex Partners: Male and female subjects who have had 1 - 5 lifetime male sex partners
- >= 6 Male Sex Partners: Male and female subjects who have had 6 or more lifetime male sex partners
Arm/Group | 0 Male Sex Partners | 1-5 Male Sex Partners | >= 6 Male Sex Partners
Number analyzed (Participants) | 82 | 13 | 5
Participants
  Responder | 78 | 13 | 1
  Non-responder | 4 | 0 | 4
Statistical Analysis 1: Comparison: 0 Male Sex Partners vs >= 6 Male Sex Partners; Test type: Superiority or Other; p = 0.0003, Univariate regression, logistic; Odds Ratio (OR) = 0.015, 95% CI 2-sided [0.00 to 0.19] — The reference group is hte "0 Partners" group
Statistical Analysis 2: Comparison: 0 Male Sex Partners vs 1-5 Male Sex Partners; Test type: Superiority or Other; p = 1.0000, Univariate regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.00 to 10.01] — The reference group is the "0 Partners" group

20. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: TOTAL LIFETIME FEMALE SEX PARTNERS
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Total number of lifetime female sex partners was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- 0 Female Sex Partners: Male and female subjects who have never had a female sex partner
- 1-5 Female Sex Partners: Male and female Subjects who have had 1 - 5 lifetime female sex partners
- >= 6 Female Sex Partners: Male and female subjects who have had 6 or more lifetime female sex partners
Arm/Group | 0 Female Sex Partners | 1-5 Female Sex Partners | >= 6 Female Sex Partners
Number analyzed (Participants) | 78 | 15 | 7
Participants
  Responder | 72 | 14 | 6
  Non-responder | 6 | 1 | 1
Statistical Analysis 1: Comparison: 0 Female Sex Partners vs >= 6 Female Sex Partners; Test type: Superiority or Other; p = 0.5503, Univariate regression, logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.05 to 4.86] — The reference group is the "0 Partners" group
Statistical Analysis 2: Comparison: 0 Female Sex Partners vs 1-5 Female Sex Partners; Test type: Superiority or Other; p = 0.8904, Univariate Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.13 to 10.46] — The reference group is the "0 Partners" group

21. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: EVER DRANK ALCOHOL
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Whether participants ever drank alcohol was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Ever Drank Alcohol: NO: Subjects who have never drank alcohol
- Ever Drank Alcohol: YES: Subjects who have drank alcohol
Arm/Group | Ever Drank Alcohol: NO | Ever Drank Alcohol: YES
Number analyzed (Participants) | 62 | 40
Participants
  Responder | 58 | 35
  Non-responder | 4 | 5
Statistical Analysis 1: Comparison: Ever Drank Alcohol: NO vs Ever Drank Alcohol: YES; Test type: Superiority or Other; p = 0.3010, Univariate regression, logistic; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.12 to 1.92] — The reference group is the "Ever drank alcohol: NO" group

22. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: EVER SMOKED MARIJUANA
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Whether participants ever smoked marijuana was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Ever Smoked Marijuana: NO: Subjects who have never smoked marijuana
- Ever Smoked Marijuana: YES: Subjects who have smoked marijuana
Arm/Group | Ever Smoked Marijuana: NO | Ever Smoked Marijuana: YES
Number analyzed (Participants) | 83 | 19
Participants
  Responder | 78 | 15
  Non-responder | 5 | 4
Statistical Analysis 1: Comparison: Ever Smoked Marijuana: NO vs Ever Smoked Marijuana: YES; Test type: Superiority or Other; p = 0.0501, Univariate regression, logistic; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.06 to 1.00] — The reference group is the "Ever smoked marijuana: NO" group

23. Secondary Outcome: Outcome Measure: Qualitative Vaccine Response to Hepatitis B Surface Antigen (Binary); Predictor: EVER USED DRUGS NOT PRESCRIBE
Description: Qualitative Vaccine Response to Hepatitis B (Hep B) Surface Antigen is defined as a "Responder" if serum a'body level is >= 10 mIU/mL and a "Non- Responder" if a serum antibody level is < 10 mIU/mL. Whether participants ever used drugs not prescribed was analyzed as a potential impact factor and was measured and examined for the association with both the presence of adequate response as well as the quantitative titer one month post 2 vaccine doses.
Time Frame: Week 28
Population: as for outcome 6
Measure: Number; unit: Participants
Groups:
- Ever Used Drugs Not Prescribed: NO: Subjects who have never used drugs that were not prescribed.
- Ever Used Drugs Not Prescribed: YES: Subjects who have used drugs that were not prescribed.
Arm/Group | Ever Used Drugs Not Prescribed: NO | Ever Used Drugs Not Prescribed: YES
Number analyzed (Participants) | 97 | 5
Participants
  Responder | 89 | 4
  Non-responder | 8 | 1
Statistical Analysis 1: Comparison: Ever Used Drugs Not Prescribed: NO vs Ever Used Drugs Not Prescribed: YES; Test type: Superiority or Other; p = 0.3846, Univariate regression, logistic; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.04 to 3.61] — The reference group is the "Ever used drugs not prescribed: NO" group

24. Secondary Outcome: Immunogenicity to Hep B 18 Months After First Immunization
Description: Persistence of protective antibody response was measured by presence or absence of 10 mIU/ml HepB surface antibody and geometric mean titer of the same antibody at Week 76
Time Frame: Week 76
Population: Participants who had a week 76 Hepatitis B antibody titer were included in this analysis.
  One subject had an a'body titer at EOS visit but did not have a'body data at week 76. Since the EOS was close to week 76, the titer from EOS was recoded as the week 76 titer.
Measure: Number; unit: Participants
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 37 | 50
Participants
  Responded (>= 10mIU/ml) | 30 | 44
  Not responded (< 10mIU/ml) | 7 | 6
Statistical Analysis 1: Comparison: Recombivax vs Twinrix; Test type: Superiority or Other; p = 0.3827, Fisher Exact
Statistical Analysis 2: Comparison: Recombivax; Test type: Superiority or Other; Responding Rate = 81.08, 95% CI 2-sided [68.84 to 92.04] — Response rate=Total number subjects responded/Total number subjects in arm
Statistical Analysis 3: Comparison: Twinrix; Test type: Superiority or Other; Responding Rate = 88.0, 95% CI 2-sided [75.69 to 95.47] — Response rate=Total number subjects responded/Total number subjects in arm

25. Secondary Outcome: Immunogenicity to Hep A in the Twinrix Arm: One Month Post 2nd Vaccination
Description: Hepatitis A antibody response in those subjects in the combined vaccine arm (Twinrix) at 1 month after the 2nd vaccination. Immunogenicity to Hepatitis is given as a positive or negative response. If the Hepatitis A serology was reactive, then the participant was considered to have a positive response; if the Hepatitis A serology was non-reactive, then the participant was considered to have a negative response.
Time Frame: Week 28
Population: The data for this analysis included those in the Twinrix arm who had week 28 hepatitis A serology results.
Measure: Number; unit: percentage of participants
Arm/Group | Twinrix
Number analyzed (Participants) | 52
percentage of participants
  POSITIVE (1 month post 2nd vaccination) | 98.08
  NEGATIVE (1 month post 2nd vaccination) | 1.92
Statistical Analysis 1: Comparison: Twinrix; Test type: Superiority or Other; Exact 95% CI — A p-value has not been entered because there is only one study arm in this analysis; Responding rate = 98.08, 95% CI 2-sided [89.74 to 99.95]

26. Secondary Outcome: Immunogenicity to Hep A in Twinrix Arm: Twelve Months Post 2nd Vaccination
Description: Hepatitis A antibody response in those subjects in the combined vaccine arm (Twinrix) at 12 months after the 2nd vaccination. Immunogenicity to Hepatitis is given as a positive or negative response.
Time Frame: Week 76
Population: Subjects in the Twinrix arm who had a Week 76 hepatitis A serology results were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Twinrix
Number analyzed (Participants) | 47
percentage of participants
  Positive (12 months post 2nd vaccination) | 91.49
  Negative (12 months post 2nd vaccination) | 8.51
Statistical Analysis 1: Comparison: Twinrix; Test type: Superiority or Other; Exact 95 % confidence interval — A p-value has not been entered because there is only one study arm in this analysis; Responding Rate = 91.49, 95% CI [79.62 to 97.63]

27. Secondary Outcome: Immunogenicity to Hep A in Twinrix Arm: Overall Response (1-month or 12-month After 2nd Vaccination)
Description: Hepatitis A antibody response in those subjects in the combined vaccine arm (Twinrix) at two time points: 1 and 12 months after the 2nd vaccination. Immunogenicity to Hepatitis is given as a positive or negative response.
Time Frame: Week 28 and Week 76
Population: Subjects in the Twinrix arm who had week 28 &/or wk 76 HepA serology results were included. For overall response analysis, if a subject was reactive at either wk 28 or wk 76, then the overall response for subject was considered "Positive". If subject was non-reactive at both wk 28and wk 76, then the overall response for subject was "Negative".
Measure: Number; unit: percentage of participants
Arm/Group | Twinrix
Number analyzed (Participants) | 53
percentage of participants
  Positive: overall | 98.11
  Negative: overall | 1.89
Statistical Analysis 1: Comparison: Twinrix; Test type: Superiority or Other; Exact 95% confidence interval — A p-value has not been entered because there is only one study arm in this analysis; Responding Rate % = 98.11, 95% CI 2-sided [89.93 to 99.95] — For overall response, if a subject is reactive at either 1-month or 12-month, then the overall response is considered "Positive". If a subject is non-reactive at both 1-month and 12-month, then the overall response for this subject is "Negative"

28. Secondary Outcome: As Treated Analysis - Adequate Antibody Response to Hep B Surface Antigen
Description: The subject was considered seroresponsive to Hepatitis B Surface Antigen if the serum antibody level was greater than or equal to 10 mIU/mL. Those who received only a single vaccination, whose second vaccination was outside of the specified time window, or other cases of protocol violations were excluded from the analysis.
Time Frame: Week 28
Population: Subjects who completed both vaccinations according to the protocol were included in the analysis (as treated analysis). Those who only had 1 vaccination,whose 2nd vaccination was outside the specified time window, or other cases of protocol violations, were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 41 | 47
percentage of participants
  Responded (>=10mIU/ml) | 85.4 | 93.6
  Not responded (< 10mIU/ml) | 14.6 | 6.4
Statistical Analysis 1: Comparison: Recombivax vs Twinrix; Test type: Superiority or Other; p = 0.2938, Fisher Exact
Statistical Analysis 2: Comparison: Recombivax; Test type: Superiority or Other; 95 % confidence interval; Responding Rate % = 85.37, 95% CI 2-sided [70.83 to 94.43]
Statistical Analysis 3: Comparison: Twinrix; Test type: Superiority or Other; 95% confidence interval; Responding Rate % = 93.62, 95% CI 2-sided [82.46 to 98.66]

29. Secondary Outcome: Assessment of Youth Understanding of Vaccine Trial and Informed Consent
Description: Assessment of understanding was measured by a questionnaire containing six questions. The summary score is the sum of correct answers from six questions.
Time Frame: Screening
Measure: Mean (Standard Deviation); unit: Number of correct answers
Arm/Group | Recombivax | Twinrix
Number analyzed (Participants) | 60 | 63
Number of correct answers | 5.18 (1.24) | 5.1 (1.32)

ADVERSE EVENTS:
Arm/Group | Recombivax | Twinrix
Serious Adverse Events (participants affected / at risk) | 2/60 | 2/63
Other Adverse Events (participants affected / at risk) | 6/60 | 4/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombivax (N=60) | Twinrix (N=63)
Asthenia (General disorders) | 1 (1) | 0 (0) — In Addition to MedDRA 6.0, WHODD 2003, 2nd quarter was used for coding.
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — WHODD 2003, 2nd quarter
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombivax (N=60) | Twinrix (N=63)
Nausea (Gastrointestinal disorders) | 1 (3) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Asthenia (General disorders) | 1 (3) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Chest Pain (General disorders) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Fatigue (General disorders) | 1 (3) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Malaise (General disorders) | 1 (3) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Pain NOS (General disorders) | 1 (2) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Dengue Fever (Infections and infestations) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Upper Respiratory Tract Infection NOS (Infections and infestations) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Femure Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Appetite Decreased N OS (Metabolism and nutrition disorders) | 1 (3) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) — WHODD 2003, 2nd quarter also used for coding
Headache (Nervous system disorders) | 5 (7) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Tremor (Nervous system disorders) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1) — WHODD 2003, 2nd quarter also used for coding
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — WHODD 2003, 2nd quarter also used for coding
Internal Fixation of Fracture (Surgical and medical procedures) | 1 (1) | 0 (0) — WHODD 2003, 2nd quarter also used for coding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.